CLINICAL TRIAL: NCT05844579
Title: ReLatIonship BEtween Implementation of Evidence-based and suppoRtive ICU cAre and ouTcomes of patIents With Acute respiratOry Distress syNdrome
Brief Title: The ICU LIBERATION Study
Acronym: LIBERATION
Status: Recruiting | Type: Observational
Sponsor: Japanese Society for Early Mobilization (Other)
Responsible Party: Sponsor
Other Study IDs: 2200115
Record Dates: First submitted 2023-04-02; First posted 2023-05-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Respiratory Distress Syndrome; Post Intensive Care Syndrome; Treatment Compliance; Quality of Life
MeSH Terms: conditions — Respiratory Distress Syndrome; postintensive care syndrome; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a condition associated with hypoxemia due to noncardiogenic causes and results in high mortality. However, the epidemiology and treatment strategy for ARDS may have changed significantly due to the accumulation of a large body of knowledge, following the two-year pandemic of the novel coronavirus (SARS-CoV-2) of which the primary manifestation is ARDS. To improve the quality of ICU care that patients receive after admission to the ICU, a variety of academic societies, including the Japanese Society of Intensive Care Medicine and the Society of Critical Care Medicine, are currently developing evidence-based guidelines and consensus guidelines and statements regarding ABCDEF bundles, nutritional therapy, ICU diary. The ABCDEF bundle, nutritional therapy, and ICU diary have been developed and are being promoted for implementation in hospitals around the world. The implementation of evidence-based ICU care is strongly recommended, especially for patients with acute respiratory distress syndrome who frequently require ventilators to maintain their lives, because their patient outcomes are worse than those who were admitted to ICU with other causes.

However, there is still little evidence on how the quality of ICU care (compliance rate) correlates with patient prognosis and outcomes, and there are currently no clear goals or indicators for the ICU care we should develop.

This study aims to investigate the epidemiology and treatments given to the patients and evaluate the implementation of evidence-based ICU care and its association with the outcomes of patients with acute respiratory distress syndrome admitted to the ICU. The contents of mechanical ventilation settings, respiratory conditions, and the evidence-based ICU care, such as analgesia, sedation, rehabilitation, and nutrition, given to the patients will be collected in a daily basis.

Aim 1: Epidemiology Aim 2: Treatments Aim 3: Evidence-based ICU care Aim 4: ARDS related Post Intensive Care Syndrome

DETAILED DESCRIPTION:
Background:

Acute respiratory distress syndrome (ARDS) is a condition associated with hypoxemia due to noncardiogenic causes with bilateral lung infiltrates on chest X-ray or CT imaging. 10% of all ICU admissions are ARDS patients, and the recent pandemic of the novel coronavirus has dramatically increased the number of ARDS patients in ICUs across the world. The international epidemiological study (2016) reported a mortality rate of 35-46% for ARDS, and this is very high mortality compared to other ICU diseases. Furthermore, ARDS survivors present with many functional impairments, including physical, cognitive, and psychiatric dysfunction (Post Intensive Care Syndrome, PICS), and their Activities of Daily Living (ADL) and Quality of Life (QOL) are impaired and many other functional impairments have been pointed out. Their inability to get their original life has attracted significant research attention and become a significantly important research topic. Many patients who are unable to return to work due to functional disability require nursing care, and there is concern about the increased burden on the patient, the family supporting the patient, and the social economy. Therefore, the development of effective strategies for patients with ARDS that take into account not only mortality but also functional prognosis is strongly needed.

Recent studies have shown that lung-protective ventilation (low tidal volume and airway pressure control), neuromuscular blocking agents, prone position, noninvasive mechanical ventilators, and extracorporeal membrane oxygenation (ECMO) have improved outcomes, including mortality, in patients with ARDS. However, the mortality of patients with ARDS is still as high as 40%. In addition, the complete reintegration ratio of patients with ARDS after 1 year of hospital discharge reported in 2003 was only 50%, and recent reports have shown little progress in this aspect. Strategies to improve outcomes (mortality and functional prognosis) of ARDS patients by improving not only treatment but also the quality of ICU care have become a hot topic in recent years. The previous paper showed that excessive sedation and absolute bed rest for the purpose of ventilation control and rest during intubation in ARDS patients correlated with delirium, prolonged duration of ventilation, and even increased mortality. Therefore, attempts have been explored to improve outcomes for ARDS patients by systematically providing sedation, analgesia, rehabilitation, spontaneous breathing and awaking tests, and delirium management during ICU admission. These attempts, known as the ABCDEF bundle, have been actively recommended by a number of academic societies to be introduced in ICUs as an attempt to improve outcomes of patients with ARDS and promote their reintegration into society. (ABCDEF bundle: A (Assess, prevent, and manage pain), B (Both spontaneous awakening trials (SAT) and spontaneous breathing trials (SBT)), C (Choice of analgesia and sedation), D (Delirium: assess, prevent, and manage), E (Early mobility and exercise), F (Family engagement and empowerment)), and even ICU care such as nutritional therapy and ICU diaries have been shown to improve outcomes for ICU patients, including ARDS, and are strongly recommended. (In this study, this ICU care is referred to as evidence-based ICU care.) On the other hand, our research team has reported that the overall implementation rate of these evidence-based ICU care, ABCDEF bundles, nutritional therapy, and ICU diaries in ICU patients is quite low, and the rate is significantly lower in mechanically ventilated patients. The reason for the low implementation rates is thought to be that the ventilator is a major barrier. Although many articles have proposed evidence-based ICU care, there is little evidence as to which of these should be prioritized and which should be combined to maximize patient outcomes. The reason for this may be that there is a lack of evidence on which of these should be prioritized and which should be combined to maximize patient outcomes. Implementation of evidence-based ICU care requires many resources and effort, and it is difficult to implement all of them simultaneously. Therefore, the purpose of this international multicenter study is to investigate the current epidemiology and treatment strategy given to the patients with ARDS after the two-year pandemic of the novel coronavirus, clarify the actual implementation of ICU care for ARDS patients who require ventilators at high frequency, and evaluate how the implementation of evidence-based ICU care is associated with patient outcomes.

Significance of the study This study has the potential to increase the generalizability of the results which will be obtained from all regions of the world, including Asia, Europe, North and South America, Oceania, and Africa. Therefore, the results will potentially contribute to improving patient treatment and outcomes in all regions of the world. Furthermore, the results obtained will provide a detailed picture of the current ICU care given to patients with ARDS in the ICU. The association/correlation analysis between its implementation and patient outcomes will identify the content of ICU care which can maximize improvement in outcomes for ARDS patients. As a result, this study will contribute to the development of ICU care guidelines and thereby improve the outcomes of patients with ARDS. The study will play a significant role in improving outcomes for patients with ARDS worldwide. In addition, the results of this study will serve as basement data for future interventional research.

ELIGIBILITY:
Inclusion Criteria:

1. Patients on an invasive or non-invasive ventilator within 24 hours of ICU admission
2. Patients who are expected to be on an invasive and/or non-invasive ventilator for more than 48 hours in total
3. Patients who meet the diagnosis of ARDS within 24 hours of ICU admission

Exclusion Criteria:

1. Patients who are younger than 16 years old
2. Patients with terminal conditions at the time of ICU admission
3. Patients who have been admitted to the ICU with a terminal care policy or who are expected to be admitted to the ICU with a terminal care policy within 24 hours of admission to the ICU
4. Patients who have expressed their refusal to have their clinical data used in research.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The following Berlin definition of ARDS will be used
  1. Acute onset (within 1 week of an apparent trigger or the appearance or worsening of respiratory symptoms)
  2. Chest imaging (plain X-ray/CT) (pleural effusion, atelectasis, bilateral shadows that cannot be explained by nodules alone)
  3. Causes of pulmonary edema (cannot be explained by cardiac insufficiency or excessive fluid infusion alone)
  4. Impaired oxygenation (PEEP/CPAP ≥ 5 cmH2O and P/F ratio < 300 mmHg)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | at the time of hospital discharge (an average of 20 days)
  For Aim 1
Compliance of lung protective ventilation defined as Tidal Volme < 6ml/kg, Plateau Pressure < 30 cmH2O, and Driving Pressure < 15cmH2O that can be measured on the mechanical ventilator | within the first two weeks of ICU admission
  For Aim 2
The implementation rate of an entire and each component of the ABCDEF bundle | within the first two weeks of ICU admission
  For Aim 3
Incidence of Post Intensive Care Syndrome | at the time of follow-up 3 months after hospital discharge
  For Aim 4: Post Intensive Care Syndrome defined as any of the following criteria; (1) physical impairment defined as the presence of Barthel Index 90 and less, (2) cognitive impairment defined as the presence of MMSE below 24 , or (3) mental health disorders defined as the presence of HADs Anxiety 8 or higher, HADs Depression 8 or higher, or IES-R 25 or higher

CONTACTS AND LOCATIONS:
Locations (1):
- LIBERATION Study Research Office, Tokyo, Japan